CLINICAL TRIAL: NCT04825353
Title: Endoscopic Combined Intrarenal Surgery for Management of Large Renal Stones: A Randomized Controlled Trial
Brief Title: Endoscopic Guided PCNL Versus Standard PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Associate professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDIRB2017122601-268
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Stones, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECIRS-Group (Experimental)
  Interventions: Procedure: Endoscopic compbined guided PCNL
- SPCNL-GRoup (Active Comparator)
  Interventions: Procedure: Standard PCNL

INTERVENTIONS:
Procedure: Endoscopic compbined guided PCNL — patient undergo stone removal by ECIRS
  Arms: ECIRS-Group
Procedure: Standard PCNL — patient undergo SPCNL
  Arms: SPCNL-GRoup

SUMMARY:
currently, percutaneous nephrolithotomy (PCNL) is the standard procedure of choice for management of large renal more than 2 cm.

the pivotal step in performing PCNL is creation of proper tract. this step can be done monitored under guidance of different modalities such as fluoroscopy, ultrasonography, endoscopy or combined in ECIRS, tract creation is controlled under endoscopic vision with a flexible ureteroscope .

DETAILED DESCRIPTION:
Aim: compare safety and efficacy and adverse events of ECIRS in comparison of standard fluoroscopic guided PCNL.

patients & methods: Patients will randomly be divided into two equal groups:

Group A: Patient will undergo ECIRS.

Group B: Patient will undergo standard PCNL

ELIGIBILITY:
Inclusion Criteria:

* patients with renal stones diameter of at least 2 cm.
* American Society of Anesthesiology score ≤ 2.

Exclusion Criteria:

* patients with renal anomalies.
* transplanted kidney.
* uncorrected coagulopathy.
* active infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Stone Free Rate | 1day after operation.
  If their is any residual stones
Stone Free Rate | 1 months post operative
  If their is any residual stones
Stone Free Rate | 3 months post-operative
  If their is any residual stones

SECONDARY OUTCOMES:
operative time | intra oprative
  the length of operation
blood loss | pre-operative and 1 day post-oprative
  hemoglobin drop

CONTACTS AND LOCATIONS:
Locations (1):
- Banha university hospital, Banhā, Qalyubia Governorate, Egypt